CLINICAL TRIAL: NCT03689998
Title: Clinical Evaluation of Topical Melatonin Application on Implant Stability of Immediate Dental Implant in Anterior & Premolar Region in Systemically Healthy Patients (Randomized Clinical Trial)
Brief Title: Evaluation of Melatonin Application of Immediate Dental Implant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed magdy Mahmoud Abdellatif, associate lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: per21085
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2020-01

CONDITIONS: Immediate Dental Implant
Keywords: immediate implant; melatonin; atrumatic extraction
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- implant placement with melatonine (Experimental): immediate implant placement with melatonine
  Interventions: Device: immediate implant placement; Drug: Melatonin
- immediate implant placement alone (Active Comparator): immediate implant placement alone
  Interventions: Device: immediate implant placement

INTERVENTIONS:
Device: immediate implant placement — immediate implant placement in freshly extraction socket
  Other Names: post extraction dental implant
Drug: Melatonin — topical application of melatonin
  Arms: implant placement with melatonine

SUMMARY:
The presence of periapical pathology, the absence of kera¬tinized tissue and lack of complete soft tissue closure over the extraction socket have been reported a drawbacks of immediate implant placement .

As mentioned before the presence of periapical pathology is one of the limitation of immediate implant placement, melatonin has an action against Gram-positive and Gram-negative microorganisms with a higher efficacy on the latter; it also showed efficacy against different strains of antibiotic-resistant bacteria.

Melatonin was found to be effective in several cases as an anxiolytic and analgesic agent. It also reduce inflammatory pain by blocking the production of nitric oxid Also the lack of complete soft tissue closure over the extraction socket is one of the drawbacks of immediate implant placement; melatonin induces the production of interleukin-1, tumor necrosis factor (TNF)-α and transforming growth factor (TGF). In addition, melatonin is an immunomodulator and a neuroendocrine hormone, and stimulates both monocyte cytokine and fibroblast proliferation, which influence angiogenesis and wound healing..

As the initial implant stability is one of the criteria of implant success, Melatonin was found to increase new cortical bone width and length during the early stages (15 and 30 days), and it also promoted early cell differentiation. Melatonin acted on the bone as a local growth factor .

DETAILED DESCRIPTION:
Melatonin is chemically recognized as N-acetyl-5-methoxytryptamine. It is a compound occurring naturally in plants, microbes and animals. The circulating level of the melatonin hormone in animals shows interesting variations, by entertainment of variable biological functions in a daily cycle "circadian rhythm". Melatonin called hormone of night is secreted by the pineal gland, and its plasma levels concentration are 50 folds higher in night in comparison to daytime. A variety of peripheral cells play a role in production of melatonin such as epithelial cells, bone marrow cells, and lymphocytes. Though melatonin is a hormone, it does not act on a specific organ, it has several functions; stimulation of the synthesis of type I collagen fibers, regulation of the body temperature, sexual development, antioxidant scavenging and detoxifying free radicals thus inhibiting the process of bone resorption through interfering with the function of osteoclasts.

ELIGIBILITY:
Inclusion criteria

1. Age: 18-60.
2. Healthy patients
3. Non Smoker
4. Patients with adequate bone volume for immediate dental implant procedure.
5. Patients with absence of any periapical pathosis.

Exclusion criteria:

1. Heavy smokers.
2. Systemic disease that contraindicates implant placement or surgical procedures.
3. No or poor patient's compliance.
4. Psychological problems.
5. Pathology at the site of intervention.
6. Pregnancy females.
7. Patient refuses to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pt. eligible for implant placement after 18 years
Enrollment: 24 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
implant stability | 6 months
  measuring implant stability using ostell

SECONDARY OUTCOMES:
Soft tissue healing | 10 days
  measuring the soft tissue healing by likert scale which classify the healing in to 5 score ( score 0 ,1 , 2 , 3 , 4 ( 0 indicate complete healing & 4 indicate incomplete healing
Post operative pain | 10 days
  measuring the post operative pain by visual analog scale from 1 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Mona Shoeib, Phd, Study Chair — Cairo University; Mona Darhous, Phd, Study Chair — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
i will check with the study chair

REFERENCES:
- [Background] El-Gammal MY, Salem AS, Anees MM, Tawfik MA. Clinical and Radiographic Evaluation of Immediate Loaded Dental Implants With Local Application of Melatonin: A Preliminary Randomized Controlled Clinical Trial. J Oral Implantol. 2016 Apr;42(2):119-25. doi: 10.1563/aaid-joi-D-14-00277. Epub 2015 Jun 23. PMID 26103559